CLINICAL TRIAL: NCT07048821
Title: The Impact of Mediterranean Diet on Patients With Hashimoto Thyroiditis
Brief Title: The Impact of Change of Thyroid Antibodies on Hormone Level and Disease Burden in Patients With Hashimoto's Thyroiditis
Acronym: Anti-TPO/TG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherihan AboElyazed Mohamed Khalil (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Sherihan AboElyazed Mohamed Khalil, Lecturer of Endocrinology and Internal Medicine Faculty of Medicine, Ain Shams University Cairo, Egypt, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS 232/2023
Record Dates: First submitted 2025-06-17; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hashimoto Thyroiditis; Mediterranean Diet
Keywords: Anti-TPO; Anti-TG; Hashimoto Thyroiditis; Mediterranean Diet; ThyPRO questionnaire
MeSH Terms: conditions — Hashimoto Disease | interventions — Diet Therapy; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with hashimoto thyroiditis (Experimental): The investigators advised patients to follow a modified Mediterranean diet plan with a reduction in goitrogenic foods for 12 weeks.
  Interventions: Dietary Supplement: Dietary modification

INTERVENTIONS:
Dietary Supplement: Dietary modification — 3-month dietary plan
  Other Names: Mediterranean diet

SUMMARY:
Hashimoto's thyroiditis (HT) is an autoimmune disease affecting the thyroid gland and is one of the most common causes of hypothyroidism. Eating habits may affect the risk of several inflammatory and immune diseases, such as HT. The current knowledge of the diet in HT is insufficient. The Mediterranean diet (MD) is an anti-inflammatory diet characterized by frequent consumption of olive oil, unrefined cereals, fresh or dried fruit and vegetables, moderate amounts of fish, dairy, and meat, and many condiments and spices. It is rich in nutrients and bioactives, which have the potential to offer anti-inflammatory aspects.

DETAILED DESCRIPTION:
The investigators aimed to assess the impact of the Mediterranean diet on patients with Hashimoto thyroiditis using the following outcomes:

Primary outcomes: Anti-TPO antibodies, Anti-Thyroglobulin antibodies, TSH, T3, T4 Secondary outcomes: BMI, Lipid profile, Symptoms of hypothyroidism

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of hypothyroidism (hypothyroid/euthyroid)
* Positive anti-thyroid antibodies (anti-TPO/anti-TG).

Exclusion Criteria:

* Pregnant or lactating females
* Age below 20 years and above 50 years
* presence of any other medical disorder

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Changes in the serum level of anti-TPO and Anti-TG antibodies | after 3 months of dietary modification
  IU/ml
Changes in the serum level of TSH | after 3 months of dietary modification
  uIU/ml
Changes in the serum level of free T3 | after 3 months of dietary modification
  pg/ml
Changes in the serum level of free T4 | after 3 months of dietary modification
  ng/dl

SECONDARY OUTCOMES:
changes in BMI | after 3 months of intervention
  kg/m^2
changes in serum level of total cholesterol, triglyceride, low-density lipoprotein, high-density lipoprotein | after 3 months of intervention
  mg/dl
Symptoms of hypothyroidism | after 3 months of intervention
  Thypro Scale

CONTACTS AND LOCATIONS:
Overall Officials: Manal Abushady, MD, Study Director — faculty of medicine, Ain Shams University
Locations (1):
- Ain Shams University hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Groenewegen KL, Mooij CF, van Trotsenburg ASP. Persisting symptoms in patients with Hashimoto's disease despite normal thyroid hormone levels: Does thyroid autoimmunity play a role? A systematic review. J Transl Autoimmun. 2021 Apr 15;4:100101. doi: 10.1016/j.jtauto.2021.100101. eCollection 2021. PMID 34027377
- [Result] Watt T, Hegedus L, Bjorner JB, Groenvold M, Bonnema SJ, Rasmussen AK, Feldt-Rasmussen U. Is Thyroid Autoimmunity per se a Determinant of Quality of Life in Patients with Autoimmune Hypothyroidism? Eur Thyroid J. 2012 Oct;1(3):186-92. doi: 10.1159/000342623. Epub 2012 Sep 29. PMID 24783018
- [Result] Watt T, Hegedus L, Groenvold M, Bjorner JB, Rasmussen AK, Bonnema SJ, Feldt-Rasmussen U. Validity and reliability of the novel thyroid-specific quality of life questionnaire, ThyPRO. Eur J Endocrinol. 2010 Jan;162(1):161-7. doi: 10.1530/EJE-09-0521. Epub 2009 Oct 1. PMID 19797502
- [Result] Danailova Y, Velikova T, Nikolaev G, Mitova Z, Shinkov A, Gagov H, Konakchieva R. Nutritional Management of Thyroiditis of Hashimoto. Int J Mol Sci. 2022 May 5;23(9):5144. doi: 10.3390/ijms23095144. PMID 35563541
- [Result] Bellastella G, Scappaticcio L, Caiazzo F, Tomasuolo M, Carotenuto R, Caputo M, Arena S, Caruso P, Maiorino MI, Esposito K. Mediterranean Diet and Thyroid: An Interesting Alliance. Nutrients. 2022 Oct 4;14(19):4130. doi: 10.3390/nu14194130. PMID 36235782

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/21/NCT07048821/Prot_SAP_000.pdf